CLINICAL TRIAL: NCT00968357
Title: A Phase 2, Multicenter, Multidose, Open-Label Study to Evaluate the Safety and Immunomodulatory Effects of SCV-07 as Monotherapy or in Combination With Ribavirin in Noncirrhotic Subjects With Genotype 1 Chronic Hepatitis C Who Have Relapsed After a Response to a Course of at Least 44 Weeks Treatment With Pegylated Interferon and Ribavirin
Brief Title: Proof-of-concept Study to Evaluate the Safety and Immunomodulatory Effects of SCV 07 as Monotherapy or in Combination With Ribavirin in Noncirrhotic Subjects With Chronic Hepatitis C Who Have Relapsed
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SciClone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SCI-SCV-HCV-P2-001; NCT00514631 (obsolete NCT alias)
Record Dates: First submitted 2009-08-27; First posted 2009-08-31 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Chronic Hepatitis C
Keywords: SCV-07; relapsers; Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — golotimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SCV-07 (Experimental): Cohort 1: SCV-07 0.1 mg/kg. Cohort 2: 1.0 mg/kg per day administered SC
  Interventions: Drug: SCV-07

INTERVENTIONS:
Drug: SCV-07 — SCV-07 dosage will remain the same throughout the study for each cohort. Monotherapy Lead-in Phase Treatment (SCV-07) for 4 weeks. Combination Treatment (SCV-07 and ribavirin) for 4 weeks, following "Lead-in Phase". Re-treatment with peg INF and RBV will be offered in the "Follow-up" to patients who in the opinion of the investigator may benefit from treatment. All patients will have a total of 3 follow-up visits for safety assessments. Women of childbearing potential will be followed up monthly for approximately up to 6 months after the "end of treatment" visit. If pregnancy occurs within the follow-up period, it needs to be followed through 8 weeks after the end of pregnancy.

SUMMARY:
SCV-07 (γ-D-glutamyl-L-tryptophan) is a new immunomodulatory compound that has been developed and patented both for composition and immunomodulatory use and is a synthetic dipeptide. The efficacy of SCV 07 in treating chronic hepatitis C virus (HCV) infection is expected to arise from the drug's ability to stimulate the T-helper 1 (Th1) type immune response and to block signal transducers and activator of transcription 3 (STAT3) mediated signaling. The purpose of this study is to determine if SCV-07 alone and/or SCV-07 in combination with ribavirin is safe and potentially effective for the treatment of genotype 1 compensated chronic hepatitis C in subjects who have relapsed after a response to a previous treatment course of at least 44 weeks with pegylated interferon and ribavirin. All subjects will receive 4 weeks of SCV-07 (Lead-in Phase), followed by 4 weeks of treatment with SCV-07 in combination with ribavirin (Combination Treatment).

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects must have compensated liver disease
* Subjects must have a history of chronic hepatitis C (genotype 1), and must be relapsers
* Subject's HCV RNA viral load must be > or = 300,000 IU/mL
* Subjects must have documentation of a liver biopsy within the last 2 years

Exclusion Criteria:

* Human immunodeficiency virus (HIV) infection or hepatitis B surface antigen (HBsAg)-positive
* Clinical evidence of cirrhosis
* Autoimmune hepatitis or other autoimmune/immune-active diseases
* Insulin-dependent diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To assess the safety of SCV-07 at 2 dose levels given as a monotherapy and to assess the immunomodulatory effects of SCV-07 given at 2 dose levels for 4 weeks and in combination with ribavirin for 4 weeks after monotherapy, respectively. | 8 weeks

SECONDARY OUTCOMES:
To assess the pharmacodynamic effects of SCV 07 and the pharmacokinetics as a monotherapy and in combination with ribavirin | 8 weeks

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - AGMG Clinical Research, Anaheim, California
  - Impact Clinical Trials, Los Angeles, California
  - A Professional Corporation, Palm Springs, California
  - Arapahoe Gastroenterology, Littleton, Colorado
  - Washington Hospital Center-MedStar Research Institute, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - University of Miami School of Medicine, Miami, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - University of Louisville, Louisville, Kentucky
  - Commonwealth Biomedical Research, LLC, Madisonville, Kentucky
  - Paul Thuluvath, Baltimore, Maryland
  - Duke University Department of Medicine, Durham, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Vanderbilt Medical Center, Nashville, Tennessee
  - Baylor College of Medicine (VAMC 15), Houston, Texas
  - Kaiser Permanente, Falls Church, Virginia

REFERENCES:
- See also: Pharmaceutical Company — http://www.sciclone.com